CLINICAL TRIAL: NCT05905172
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Entecavir-based, Phase IIIb Clinical Trial of Hydronidone Capsule in the Treatment of Liver Fibrosis Associated With Chronic Hepatitis B
Brief Title: Hydronidone Capsules in Long-term Treatment in Patients With Chronic Viral Hepatitis B Liver Fibrosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDN-F351-202201
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — hydronidone; 5-methyl-1-(4-hydroxylphenyl)-2-(1H)-pyridone

STUDY DESIGN:
Intervention Model Description: Test group: hydronidone capsules, three times a day, 3 capsules each time，oral，daily therapeutic dose of 270 mg, half an hour before the meal
  Control group: placebo capsules, three times a day, 3 capsules each time，oral，half an hour before the meal.
  Basic treatment: Both test and control groups were treated with entecavir antiviral therapy, once daily, 0.5 mg per time, oral.
  In case of drug resistance or other conditions requiring dose adjustment, the investigator may adjust the dose and type of basic treatment drug appropriately.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the clinical trial begins, the test drug and placebo are packaged in the same way, and the drug number is marked on the packaging according to the random table. The subjects take the drugs according to the randomly assigned drug number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydronidone group (Experimental): Patients were given three capsules of hydronidone three times a day for 5 years.
  Interventions: Drug: Hydronidone capsules
- The placebo group (Placebo Comparator): Patients were given three capsules of placebo three times a day for 5 years.
  Interventions: Drug: The placebo capsules

INTERVENTIONS:
Drug: Hydronidone capsules — After randomization, the experimental group received hydronidone capsules three times a day, 3 capsules each time, for 5 years.
  Other Names: F351
  Arms: Hydronidone group
Drug: The placebo capsules — After randomization, The control group received three placebo capsules three times a day. 3 capsules each time, for 5 years.
  Other Names: N
  Arms: The placebo group

SUMMARY:
This study is a Phase IIIb extension trial following the "A Randomized, Double-blind, Placebo-controlled, Multicenter, Entecavir-based, Phase III Clinical Trial of Hydronidone Capsule in the Treatment of Liver Fibrosis Associated with Chronic Hepatitis B".

The main objective of this study is to evaluate the effectiveness and the safety of hydronidone capsules for long-term treatment of patients with chronic viral hepatitis B liver fibrosis.

DETAILED DESCRIPTION:
Nowadays, there is no satisfactory treatment and drug for liver fibrosis, so the etiology treatment of liver fibrosis and cirrhosis is the most important treatment. However, the etiology and treatment can not completely prevent the progression of liver fibrosis, and liver cirrhosis and liver cancer still occur after antiviral treatment. Although some drugs in domestic and foreign clinical trials have reported the effect of treating liver fibrosis, there is no recognized effective chemical drugs or biological agents against liver fibrosis. According to the available evidence, hydronidone capsules can effectively reduce the severity of liver fibrosis, which is expected to further reduce the risk of clinical endpoint events. Since the clinical benefit from the improvement of liver fibrosis usually takes a long time to observe, this trial takes an extended treatment approach to continuously evaluate the clinical benefit of subjects undergoing long-term treatment with hydronidone capsules in patients with liver fibrosis.

This study is a Phase IIIb extension trial following the "A Randomized, Double-blind, Placebo-controlled, Multicenter, Entecavir-based, Phase III Clinical Trial of Hydronidone Capsule in the Treatment of Liver Fibrosis Associated with Chronic Hepatitis B". Subjects who have completed the Phase III, placebo-controlled design, double-blind, can enter the study and continue treatment according to the original treatment protocol.The aim is to evaluate the effectiveness and the safety of hydronidone capsules for long-term treatment of patients with chronic viral hepatitis B liver fibrosis.

The test group received hydronidone capsules three times a day at a daily dose of 270 mg and oral medication half an hour before the meal. The control group received placebo capsules three times a day, half an hour before the meal.Both the test and control groups received entecavir antiviral therapy as basic treatment, once daily at 0.5 mg each, by fasting oral administration. If the subject is not suitable for entecavir, the investigator will decide on the corresponding antiviral treatment according to the subject's specific condition. Discontinuation criteria for entecavir: According to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2019 edition), the American Association for the Study of Liver Disease (AASLD) and the European Association for Liver Disease (EASL) management guidelines.

Visit examination items: clinical laboratory tests (routine ALT) every 6 months (for ALT and AST, additional tests as appropriate), HBVDNA, hepatitis B, transient elastography examination, etc. In order to improve subject compliance, the investigator may increase or reduce the examination frequency or items, and at least 1 year to reducing the frequency. Additional according to the actual situation

ELIGIBILITY:
Inclusion Criteria:

* Participate in the Phase III trial of this project (Protocol Number: KDN-F351- 202101 ，ClinicalTrials.gov ID: NCT05115942 ), complete the main treatment course and the last visit;
* Before the trial, the subject understood the nature, significance, possible benefits, possible inconvenience and potential dangers of the trial, volunteered to participate in the clinical trial, was able to communicate well with the investigator, comply with the requirements of the whole study, and signed a written informed consent.

Exclusion Criteria:

* One of any clinical endpoints occurred during the phase III trial (Note: for non cirrhotic patients, Clinical endpoints include progression to cirrhosis,decompensated cirrhosis complications [ascites, esophagogastric vein rupture and bleeding, spontaneous bacterial peritonitis, hepatorenal syndrome, hepatopulmonary syndrome, hepatic encephalopathy, portal vein thrombosis and cirrhotic cardiomyopathy], hepatocellular carcinoma, liver transplantation or liver disease related death / all-cause death; For patients with liver cirrhosis, Clinical endpoints include complications of decompensated cirrhosis, hepatocellular carcinoma, liver transplantation, or liver disease-related death / all-cause death);
* Patients with malignant tumors other than hepatocellular carcinoma and with an expected survival period of less than 1 year;
* Any opinion of the investigator that may affect the subject to provide informed consent or follow the trial protocol, or participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinical endpoint events (defined as the occurrence of any clinical endpoint event). | 5years
  For non-cirrhotic patients, clinical endpoints include progression to cirrhosis, decompensated cirrhosis complications [ascites, esophagogastric vein rupture and bleeding, spontaneous bacterial peritonitis, hepatorenal syndrome, hepatic encephalopathy, portal vein thrombosis and cirrhotic cardiomyopathy, etc.], hepatocellular carcinoma, liver transplantation or liver disease-related death / all-cause death; for patients with cirrhosis, clinical endpoints include occurrence of decompensated cirrhosis complications, hepatocellular carcinoma, liver transplantation or liver disease-related death or all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Lungen Lu, Dr, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Jun Cheng, Dr, Principal Investigator — Beijing Ditan Hospital
Locations (23):
- China (23):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Shanghai General Hospital,Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Beijing youan hospital, the capital of the capital, Beijing
  - Tsinghua Changgeng Hospital, Beijing, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The Second Xiangya Hospital, Central South University, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Three Gorges Hospital affiliated to Chongqing University, Chongqing
  - Guizhou Provincial People's Hospital, Guizhou
  - Hangzhou Xixi Hospital (Hangzhou Sixth People's Hospital), Hangzhou
  - Henan Provincial People's Hospital, Henan
  - Affiliated Hospital of Traditional Chinese Medicine of Southwest Medical University, Luzhou
  - Nanchang Ninth Hospital (Nanchang Central Hospital), Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Shenzhen Third People's Hospital, Shenzhen
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang
  - Yanbian University Affiliated Hospital, Yanbian
  - Zhenjiang Third People's Hospita, Zhenjiang
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No